CLINICAL TRIAL: NCT06193226
Title: Is Cryotherapy Effective as a Therapeutic Option for Oral Lesion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Wessam Ibrahim Shehab, Lecturer of Oral Medicine and Periodontology Department, Faculty of Dentistry, October 6 University, Egypt, October 6 University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RECO6U/11-2023
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Cryotherapy; Oral Lesions
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cryotherapy (Experimental): Cryotherapy can be done in two ways:
  1. Open technique: Using cotton swabs or a cryogun spray, the cryogen is delivered directly to the lesion in this technique.
  2. Closed technique: Cryo-probes are used to apply the cryogen to the lesion in this procedure.
  Interventions: Other: Cryotherapy

INTERVENTIONS:
Other: Cryotherapy — Cryotherapy can be done in two ways:
  1. Open technique: Using cotton swabs or a cryogun spray, the cryogen is delivered directly to the lesion in this technique.
  2. Closed technique: Cryo-probes are used to apply the cryogen to the lesion in this procedure.
  The spray's nozzle of the Cryogun spray -50 ◦C was situated 1 cm away from the skin's surface and applied on the oral lesion for 30 seconds. Each freezing cycle lasted 10 to 30 seconds, with the subsequent 60-second thaw interval lasting twice as long as the freezing time. The ice ball that formed during freezing was totally melted before the subsequent freezing process could begin.
  The application process should went from the core out to the edges. The management of lesions that are too big to be frozen by a single spray requires many overlapping treatments of liquid nitrogen. Mucoceles and erosive lichen planus took 30 to 50 seconds to freeze, whereas fibromas and leukoplakia took 60 to 70 seconds.

SUMMARY:
The aim of this study is to evaluate the effectiveness of cryotherapy as a therapeutic option for oral lesions.

DETAILED DESCRIPTION:
Low-temperature applications were originally employed by the Egyptians to treat pain, and subsequently during the Franco-Prussian War for severed limbs. Hippocrates advocated the application of cold to lessen bruising, bleeding, and discomfort, while John Hunter wrote in 1777 that "the local tissue response to freezing includes local tissue necrosis, vascular stasis, and excellent healing." Using a solution of salt and ice, James Arnott (1851) was the first to describe and demonstrate this freezing technique for malignant breast tumors.

The term "cryotherapy" was used in 1908 to describe the use of extremely low temperatures to cure skin lesions. Currently, cryotherapy involves cooling the body's surface without destroying tissue, whereas in cryosurgery, sick tissues are frozen to death.

In the technique, several cryogens include: liquid nitroglycerine (-196 °C), Nitrous oxide (0°C), Solid CO2 (-78o C), Chlorodifluoromethane (-41°C), Dimethyl ether (-24 °C) and propane (-42 °C).

The intralesional technique, open method, or closed method can all be used to apply cryogens. The best application approach for big superficial cutaneous lesions is an open spray technique, in which the spray's nozzle is situated 1 cm away from the skin's surface, and the lesion is destroyed using either a paintbrush technique or a spiral technique.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Both sexes.
* Patients who had benign intraoral epithelial lesions free of infection.

Exclusion Criteria:

* Patients with Reynaud's illness.
* Cold sensitivity.
* History of diabetes.
* Severe infections.
* Patients who had cryoglobulinemia.
* Cold urticaria.
* Patients who was receiving hemodialysis.
* Patients who was receiving immunosuppressive medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
The degree of pain | 21st days postoperatively
  The degree of pain was assessed by using Visual Analogue Scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable"), which was documented on the 1st, 3rd, 7th, 21st days after the procedure

SECONDARY OUTCOMES:
Epithelization of the lesion | 1st month postoperatively
  Number of Participants with epithelization of the lesion was evaluated in the 1st postoperative month
The incidence of recurrence of the lesion | 2nd month postoperatively
  Recurrence of the lesion was evaluated in the 2nd postoperative month

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.